CLINICAL TRIAL: NCT02879240
Title: Effectiveness of Animated Cartoons for Improving Cooperation During the Delivery of Inhaled Treatments to Young Children With Asthma
Brief Title: Animated Cartoons and Cooperation in Young Children Receiving Inhaled Medications
Acronym: DISTRACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Principal Investigator, David Drummond, M.D., Hôpital Necker-Enfants Malades
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Distract01
Record Dates: First submitted 2016-08-16; First posted 2016-08-25 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Patient Compliance; Inhalation Spacers
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group animated cartoon-black screen (AB) (Other): In this group, children will be exposed to a animated cartoon during the delivery of their inhaled treatment twice a day during one week, then they will be exposed to a black screen in the same conditions for one other week.
  Interventions: Other: Animated Cartoon; Other: Black screen
- Group black screen - animated cartoon (BA) (Other): In this group, children will be exposed to a black screen during the delivery of their inhaled treatment twice a day during one week, then they will be exposed to an animated cartoon in the same conditions for one other week.
  Interventions: Other: Animated Cartoon; Other: Black screen

INTERVENTIONS:
Other: Animated Cartoon — An animated cartoon chosen by the parents is displayed on a smartphone attached on the spacer of the child.
Other: Black screen — A video displaying a black screen is used as control, and displayed on a smartphone attached on the spacer of the child.

SUMMARY:
Up to 50% of infants and young children cry during the administration of their inhaled treatment for their asthma. This results in decreased lung deposition, and thus decreased effectiveness of their inhaled treatment.

The objective of this study is to evaluate whether animated cartoons can increase the cooperation of young children with asthma who are not cooperative during the delivery of their ICS therapy through a pMDI/spacer.

ELIGIBILITY:
Inclusion Criteria:

* Dyad parent-child.
* Parent must be 18 years or older and own a smartphone which can record videos and display animated cartoons.
* Child must be 6-47 months old, and require an inhaled corticosteroid therapy, and use a pressurized metered-dose inhaler and a spacer, and have difficulties in cooperation at least half of the time on the last week.

Exclusion Criteria:

* Children with a medical history of epilepsy, or visual or hearing impairment not corrected by an appropriate device/treatment.
* Parents not speaking French or English.
* Parents not able to run the mobile application used to record the videos of the child despite repeated explanations.

Ages: 6 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2016-08; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Fraction of time during which the child is non-cooperative | At the end of the three weeks (day 21)
  Length of time during which the child is crying or moving outside the mask, divided by the total length of time needed for the delivery of the inhaled treatment

SECONDARY OUTCOMES:
Fraction of time during which the child is crying | At the end of the three weeks (day 21)
  Length of time during which the child is crying divided by the total length of time needed for the delivery of the inhaled treatment
Fraction of time during which the child is moving outside the mask | At the end of the three weeks (day 21)
  Length of time during which the child is moving outside the mask divided by the total length of time needed for the delivery of the inhaled treatment

OTHER OUTCOMES:
Hetero-evaluation of the cooperation of the child by the parent | At the end of the three weeks (day 21)

CONTACTS AND LOCATIONS:
Overall Officials: David Drummond, M.D., Principal Investigator — Necker hospital
Locations (3):
- France (3):
  - Department of pediatrics, Mignot Hospital, Le Chesnay
  - Department of pediatric pulmonology, Hopital Robert Debré, Paris
  - Department of pediatric pulmonology, Necker Hospital, Paris

REFERENCES:
- [Background] Guilbert TW, Morgan WJ, Zeiger RS, Mauger DT, Boehmer SJ, Szefler SJ, Bacharier LB, Lemanske RF Jr, Strunk RC, Allen DB, Bloomberg GR, Heldt G, Krawiec M, Larsen G, Liu AH, Chinchilli VM, Sorkness CA, Taussig LM, Martinez FD. Long-term inhaled corticosteroids in preschool children at high risk for asthma. N Engl J Med. 2006 May 11;354(19):1985-97. doi: 10.1056/NEJMoa051378. PMID 16687711
- [Background] Iles R, Lister P, Edmunds AT. Crying significantly reduces absorption of aerosolised drug in infants. Arch Dis Child. 1999 Aug;81(2):163-5. doi: 10.1136/adc.81.2.163. PMID 10490528
- [Background] Lee J, Lee J, Lim H, Son JS, Lee JR, Kim DC, Ko S. Cartoon distraction alleviates anxiety in children during induction of anesthesia. Anesth Analg. 2012 Nov;115(5):1168-73. doi: 10.1213/ANE.0b013e31824fb469. Epub 2012 Sep 25. PMID 23011563